CLINICAL TRIAL: NCT05241249
Title: Phase II, Neoadjuvant Study of Parasympathetic Stimulation With Bethanechol in Combination With Gemcitabine and Nab-paclitaxel in Borderline Resectable Pancreatic Adenocarcinoma
Brief Title: Stimulation With Bethanechol in Combination With Gemcitabine and Nab-paclitaxel in Pancreatic Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Susan E. Bates (Other)
Responsible Party: Sponsor-Investigator, Susan E. Bates, Associate Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAT5285
Record Dates: First submitted 2022-02-03; First posted 2022-02-15 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Pancreas Cancer
Keywords: Pancreas; pancreatic adenocarcinoma; adenocarcinoma; bethanechol; parasympathetic
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — Bethanechol; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: This is a Phase IIA study evaluating short term parasympathetic activation with fixed dose bethanechol in subjects with pancreatic cancer who should proceed to surgery after 4 -6 months of chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bethanechol (Experimental): Patients with borderline resectable pancreatic cancer and no contraindication to bethanechol therapy will receive bethanechol on day 1 and continue until 2 days prior to scheduled surgery for a minimum of 2 months.
  Interventions: Drug: Bethanechol; Drug: Gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: Bethanechol — Study Drug: Bethanechol (generic), supplied as 50mg oral tablets. Subjects will take 2 tablets (100mg) twice daily. Medication should be taken 1 hour before meals in AM and PM. Medication will be purchased commercially and dispensed at the research pharmacy.
  Other Names: Bethanechol chloride tablet
Drug: Gemcitabine — Non-experimental. Chemotherapy will be administered on a day 1, 8 and 15 schedule with gemcitabine at a dose of 1000 mg/m2
Drug: nab-paclitaxel — Non-experimental. Chemotherapy will be administered on a day 1, 8 and 15 schedule with nab-paclitaxel dose at 125 mg/m2

SUMMARY:
The primary objective of this study is to assess the impact of bethanechol therapy on R0 resection rates. The safety objective will be assessment of the safety and tolerability of bethanechol in combination with gemcitabine and nab-paclitaxel. The exploratory objective will be to evaluate genomic biomarkers associated with parasympathetic stimulation in pancreatic cancer, and the ability to reduce tumor growth rate.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the drug, bethanechol, could potentially be used in combination with chemotherapy regimen gemcitabine and nab-paclitaxel and surgery to decrease the chance of the cancer coming back after it is removed. Animal models have shown that treatment with bethanechol can inhibit cancer growth and spread. The chemotherapy regimen nab-paclitaxel for use in combination with gemcitabine to treat patients with metastatic pancreatic cancer is FDA approved. Although bethanechol is FDA approved, in this study its use is experimental. The aim of the study is to show that the medication is easy to tolerate and that it shows signs of slowing cancer cell growth. The investigators hypothesize that treatment with bethanechol will alter nerve conduction within tumors by stimulating the parasympathetic nervous system and reduce tumor proliferation, decrease CD44+ expression in cancer cells, decrease tumor growth rate resulting in an improved R0 resection rate.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic Ductal Adenocarcinoma
* Plan for neoadjuvant chemotherapy
* Available diagnostic tissue adequate for biomarker analysis
* Ability to tolerate PO meds and comply with study procedures

Exclusion Criteria:

* Metastatic disease
* Evidence of GI obstruction
* Baseline bradycardia (HR<55) or hypotension (systolic blood pressure<90)
* Use of acetylcholinesterase inhibitors
* Medical conditions including: hyperthyroidism, active/symptomatic coronary artery disease, seizure disorder, peptic ulcer disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 36 months
  This rate will be analyzed in patients treated with bethanechol in combination with gemcitabine and nab-paclitaxel compared to historical R0 resection rates.

SECONDARY OUTCOMES:
Ki-67 expression in tumor cells | 36 months
  This is to measure cell proliferation by Ki-67 expression in tumor cells, to quantify the change in tumor growth and alterations in inflammatory cytokines and immune profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Bates, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No